CLINICAL TRIAL: NCT05780762
Title: Impact of an Intervention Integrating the MPHS Nursing Model of Care on the Partnership in Health, With the Patient Followed in Primary Care by an Advanced Practice Nurse (APN) for One or More Stabilized Chronic Pathologies
Acronym: IMPACT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Collaborators: Ministry of Health, France (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 21GI262; ANSM (Other: 2022-A02513-40)
Record Dates: First submitted 2022-12-05; First posted 2023-03-23 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-11

CONDITIONS: Chronic Disease
Keywords: advanced practice nurse (APN); patient partnership; health literacy; self-management
MeSH Terms: conditions — Chronic Disease

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- IMPACT program - experimental group (Experimental): patients followed for one or more stabilized chronic pathologies and benefiting from usual care with an Advanced Practice Nurse AND benefiting from the IMPACT program, which combines management at 3 levels: (1) co-definition of the health situation, (2) co-planning of care and co-actions, and (3) co-assessment with the patient and his or her care team, and incorporates evidence-based measurement tools.
  Interventions: Other: IMPACT Program
- Usal care : control group (Sham Comparator): patients followed for one or several stabilized chronic pathology(ies) and benefiting from a usual management with a Nurse in Advanced Practice.
  Interventions: Other: usal care

INTERVENTIONS:
Other: IMPACT Program — care at 3 levels:
  (1) co-definition of the health situation, (2) co-planning of care and co-actions, and (3) co-assessment with the patient and with the team caring for him or her, and incorporating evidence-based measurement tools.
  Arms: IMPACT program - experimental group
Other: usal care — usual management with a Nurse in Advanced Practice.
  Arms: Usal care : control group

SUMMARY:
The WHO and our governance advocate that health professionals should organize care around the patient, considering his or her values, needs and preferences, and enabling the patient to develop the capacity to self-manage the chronic health problems he or she faces. Chronic disease is an ongoing dynamic process and adaptation to this process is complicated by the interaction of several determinants: self-management capacity, level of health literacy, quality of life and experience of care. To best support chronic disease, the recommendation is to adopt a management strategy that allows chronic patients to play an active role in the management of their condition and in the day-to-day decision-making process. The management of chronic pathologies is one of the specialties in which Advanced Practice Nurses are positioned, in primary care, outside hospital. Nursing care benefits from care models that allow for more adapted responses, regarding particular care situations, or certain patient typologies. The Humanistic Partnership Health Care Model (MPHS) implement in current Advanced Practice Nurse (APN) practice.

DETAILED DESCRIPTION:
The IMPACT program proposes to integrate the MPHS model into primary care, within advanced practice nursing care, to strengthen the partnership of the patient with chronic disease. This model will allow the advanced practice nurse to co-construct with the patient partner a care trajectory that will be integrative, considering his aspirations and priorities to carry out his life project, while coping with his chronic pathology(ies). To do this, particular attention to the determinants of adaptation to chronic disease: self-management capacity, health literacy, quality of life and experience of care is pay.

The IMPACT program will use the theoretical framework of the MPHS model of care to structure the advanced practice nursing care management and will incorporate validated measurement tools to address the determinants of patient adaptation to chronic disease. The specific management of the IMPACT program will consist of 3 phases: (1) co-definition of the health situation, (2) co-planning of care and co-actions, and (3) co-assessment with the patient and the team caring for him/her.

ELIGIBILITY:
Inclusion Criteria:

* Followed by APN, within the framework of an organizational protocol established with a patient's referring physician, for the management of one or more chronic pathology(ies) from the following list: stroke; chronic arterial disease; heart disease, coronary artery disease; type 1 diabetes and type 2 diabetes; chronic respiratory failure; Parkinson's disease; epilepsy
* Affiliated or entitled to a social security plan
* Having received informed information about the study and having co-signed, with the investigator, a consent to participate in the study

Exclusion Criteria:

- Patient not referred by a physician for APN follow-up

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 420 (Estimated)
Dates: Start 2024-04-12 (Actual); Primary Completion 2028-02-28 (Estimated); Study Completion 2028-11-30 (Estimated)

PRIMARY OUTCOMES:
The patient/advanced practice nurse partnership | At month 9
  The patient/advanced practice nurse partnership will be assessed by a measure via the PIH-Fv (Partners In Health scale French version) questionnaire at 9 months.
  The PIH-Fv (Partners In Health scale in French version) questionnaire was developed and validated in French by Hudon et al. The PIH-Fv scale is a self-assessment questionnaire that includes 12 items, which are answered using 9-point Likert-type scales. The total score goes from 0 to 96: 0 representing poor self-management and 96 better self-management.

SECONDARY OUTCOMES:
The patient/advanced practice nurse partnership across the continuum of care | baseline, 3 and 6 months
  Measurement of the impact of the intervention on the partnership via the Partners In Health scale French version.This questionnaire is a self-assessment questionnaire that includes 12 items, which are answered using 9-point Likert-type scales. The total score goes from 0 to 96: 0 representing poor self-management and 96 better self-management.
Perception of health-related quality of life | At inclusion, 3, 6 and 9 months.
  Measurement of the perception of health-related quality of life via the World Health Organisation Quality Of Life questionnaire. This questionnaire questions 4 domains: physical health, psychological health, social sphere and environment. The patient answers according to 3 groups of 5 modalities of the Likert scale. The first group goes from " very weak " to " very good"; the second goes from " very unsatisfied " to "very satisfied" ; the third goes from "not at all" to " extremely"
Health literacy level | at inclusion, 3, 6 and 9 months
  Measurement of health literacy level via the European Health Literacy Survey (HLS-EU16) questionnaire validated in French version. It consists of 16 items, for which the patient answers according 4 modalities "very easy" to "very difficult".
Impact of the quality of advanced practice nurse consultation from patient's perspective | At baseline, 3, 6 and 9 months
  Measurement of the impact of the advanced practice nurse consultation on the patient's perceived ability to understand and cope with his or her health problems and illness via the PEI questionnaire vf (Patient Enablement Instrument French version) questionnaire. It consists of 6 questions to which the patient responds in 3 ways "much more", "more", or "as before the visit or less"
Adoption of IMPACT program by advanced practice nurse | 3 years
  Adoption of IMPACT program by advanced practice nurse will be assessed by number of advanced practice nurses including patients and number of patients followed by each APN
Participation in IMPACT program | 3 years
  Participation in IMPACT program will be assessed by number of patients who agreed to be followed with this model of care/number of patients who were offered follow-up
IMPACT program satisfaction for advanced practice nurse | 3 years
  IMPACT program satisfaction will be assessed by semi-structured interview with advanced practice nurse
effectiveness of IMPACT program | 3 years
  Effectiveness of IMPACT program will be assessed by proportion of patients completing the proposed follow-up package
Context of IMPACT program | 3 years
  Context of IMPACT program will be assessed with semi-structured interviews with advanced practice nurse which will evaluate factors favoring and hindering the implementation, the adaptation, the achievement and sustainbility of the IMPACT program

CONTACTS AND LOCATIONS:
Overall Officials: Elise VEROT, MD, Principal Investigator — CHUSE
Locations (5):
- France (5):
  - CH le Corbusier - Firminy, Firminy
  - Hôpital du Gier, Saint-Chamond
  - Centre Hospitalier Universitaire - Pneumologie, Saint-Etienne
  - Centre Hospitalier Universitaire - Cardiologie, Saint-Etienne
  - Direction de la Prévention et de la Santé des Populations, Saint-Etienne

IPD SHARING:
Plan to Share IPD: No